CLINICAL TRIAL: NCT00659347
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study of DOV 21,947 in Patients With Major Depressive Disorder
Brief Title: Efficacy and Safety of DOV 21,947 in the Treatment of Major Depressive Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: DOV Pharmaceutical, Inc. (Industry)
Responsible Party: Dr. Nuoyo Huang, Vice President Clinical Research and Development, DOV Pharmaceutical, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DOV 947-010
Record Dates: First submitted 2008-04-09; First posted 2008-04-16 (Estimated); Last update posted 2008-12-05 (Estimated); Status verified 2008-12

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: DOV 21, 947
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DOV 21, 947 — Capsules, 25 mg, 2 capsules (1 Active/1 Placebo) BID, 2 weeks Capsules, 25 mg, 2 capsules (2 Active) BID, 2 weeks
  Arms: 1
Drug: Placebo — Capsules,25 mg,BID,6weeks
  Arms: 2

SUMMARY:
The primary objectives of this placebo-controlled trial are to evaluate effectiveness and safety of DOV 21,947 at two oral dose levels.

DETAILED DESCRIPTION:
DOV 21,947 is an investigational drug that is being developed for the treatment of depression. The purpose of this study is to evaluate the safety and effectiveness of a flexible dosing schedule of DOV 21,947 (25 mg twice daily for two weeks, then 50 mg twice daily for four weeks as compared to placebo) in the treatment of major depressive disorder. Information about any side effects that may occur will also be collected.

The efficacy evaluation will be based on the change in the total MADRS and HAMD-17 scores from randomization to week 9 .The secondary objective is to determine if DOV 21,947 improves the quality of life for patients with MDD as compared to placebo

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between 18 and 65 years of age (inclusive).
2. Either outpatients or inpatients diagnosed with major depressive disorder (MDD) according to Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR, see Appendix 3) and MINI International Neuropsychiatric Interview (MINI).
3. Patients with recurrent depressive episode of at least 2 months in duration. Patients must have previously responded (significant clinical improvement judged by the Principal Investigator) to at least one antidepressant treatment.
4. HAMD-17 total score * 22 with a severity score of at least 2 on Item 1 at the Placebo Run-In Visit and the Baseline/Day 1 Visit.
5. HAMD-17 score reduction ≤ 15% between the Placebo Run-In Visit and the Baseline/Day 1 Visit.
6. HAM-A total score < 17 at the Screening Visit.

Exclusion Criteria:

1. Patients with a HAMD-17 total score reduction of more than 15% between the Placebo Run-In Visit and the Baseline/Day 1 Visit (placebo responders).
2. Patients with a medical history of MDD that consistently did not respond significantly to an adequate treatment regimen of a monoamine oxidase (MAO) inhibitor.
3. Patients who are known to be antidepressant treatment-resistant. Patients are defined as treatment-resistant if in the past they have failed adequate antidepressant treatments (dose level approved in the product labeling and was administered for at least 4 weeks) from two or more different pharmacological classes (e.g., TCA, SSRI, SNRI, MAO-I, etc). Failure to respond to an adequate antidepressant treatment is defined as the absence of at least a 50% improvement in symptoms by patient report or documented history, or lack of significant clinical improvement at the Principal Investigator's discretion.
4. Patients with a medical history of MDD who consistently did not respond significantly to electroconvulsive shock therapy (ECT) or had ECT within a year prior to the Screening Visit regardless of outcome.
5. Patients with psychotic depression

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be the change in tot al score of MADRS scale. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nuoyu Huang, MD/PhD, Study Director — DOV Pharmaceutical, Inc.
Locations (26):
- United States (10):
  - Comprehensive Psychiatric Care, Norwich, Connecticut
  - Future Care Studies, Springfield, Massachusetts
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - CRI Worldwide, LLC, Clementon, New Jersey
  - Princeton Medical Institute, Princeton, New Jersey
  - Brooklyn Medical Institute, Brooklyn, New York
  - Social Psychiatry Research Institute, New York, New York
  - Richmond Behavorial Associates, Staten Island, New York
  - CRI Worldwide, LLC, Philadelphia, Pennsylvania
  - Scranton Medical Institutes, Scranton, Pennsylvania
- Romania (12):
  - Spitalul Judetean Arges, Piteşti, Argeş
  - Spitalul Clinic de Neurologie si Psihiatrie Oradea, Oradea, Bihor County
  - SC Corpores Sana Medical SRL, Bucharest, Bucharest
  - Spitalul Clinic "Colentina", Ambulator Specialitate, Sectia Psihiatrie, Bucharest, Bucharest
  - Spitalul Clinic de Psihiatrie "Prof. Dr. Alexandru Obregia", pavilion III, Bucharest, Bucharest
  - Spitalul Clinic de Psihiatrie "Prof. Dr. Alexandru Obregia", Pavilion IV, Bucharest, Bucharest
  - Spitalul Clinic de Psihiatrie "Prof. Dr. Alexandru Obregia", Pavilion X, Bucharest, Bucharest
  - Cabinetul Medical Lorentina 2102 S.R.L., Târgovişte, Dâmbovița County
  - Spitalul Clinic de Psihiatrie "Socola", Lasi, Lasi
  - Spitalul Judetean de Urgenta Piatra Neamt, Piatra Neamţ, Piatra Neamt
  - Spitalul Clinic Judetean de Urgenta Targu Mures, Târgu Mureş, Targu Mures
  - Spitalul Universitar de Psihiatrie "Socola", Lasi
- Serbia (4):
  - Institut za mentalno zdravlje Palmoticeva 37, Belgrade
  - Institut za psihijatriju KCS, Belgrade
  - Klinika za neurologiju i psihijatriju, Kragujevac
  - Klinika za psihijatriju Vojnomedicinske Akademije, Velgrade